CLINICAL TRIAL: NCT06622772
Title: Evaluation of a Novel Valsalva Assist Device for Terminating Supraventricular Tachycardia: a Randomized Controlled Trial
Brief Title: A Novel Valsalva Assist Device for Terminating Supraventricular Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Songnan Li, Chief physician, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS2023109
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Supraventricular Tachycardia (SVT)
Keywords: supraventricular tachycardia; Valsalva Manoeuvre
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Masking Description: All analyses were done by statisticians masked to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VAD group (Experimental): Valsalva manoeuvre with a valsalva assist device (VAD)
  Interventions: Device: Valsalva assist device
- Control group (Other): standard Valsalva manoeuvre
  Interventions: Other: standard Valsalva manoeuvre

INTERVENTIONS:
Device: Valsalva assist device — A valsalva assist device designed to provide the recommended resistance to exhalation at a pressure of 40 mmHg.
  Arms: VAD group
Other: standard Valsalva manoeuvre — The Valsalva manoeuvre is carried out without any device.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate the efficiency of a device for terminating supraventricular tachycardia. The main questions it aims to answer are:

The Valsalva manoeuvre is a first-line treatment for supraventricular tachycardia, but the success rate is low. Can the device help to increase the sucess rate? Whether the device is effective and safe to use at home? Researchers will compare whether the device is more effective than a standard Valsalva manoeuvre to treat supraventricular tachycardia.

Participants will:

be randomly assigned (1:1) to a standard Valsalva manoeuvre group (control) or Valsalva manoeuvre with the device (intervention) .

DETAILED DESCRIPTION:
- Quality control and quality assurance: Over the first month of the trial, clinical investigators will come off-line for active participation once all local regulatory requirements have been met. Training for Valsalva manoeuvre procedure, data collection and reporting must be completed. Endpoint and Adverse Event Committee will be installed comprising of medical experts who are not involved in the study.

Periodic monitoring visits will be made throughout the clinical study to assure that the Investigator obligations are fulfilled, and all applicable regulations and guidelines are being followed. Key variables (demographics, inclusion/exclusion criteria, and safety) on the CRFs will be compared with each subject's source documents. Any discrepancies will be noted and resolved.

The auditor will check potential problems, evaluating whether their study implementation, data collection and data analysis are in accordance with the protocol, Manual of procedure (MOP) and good clinical practice (GCP) guidelines. CRFs, source documents and other study files must be accessible at all study sites at the time of auditing and inspection during the course of the study and after the completion of the study.

- Sample size: To calculate the required sample size, we estimated that the standard Valsalva manoeuvre would cause cardioversion in 20% of patients with supraventricular tachycardia on the basis of local audit data and previous studies. In our pro-protocol study, 40 patients were included, and the conversion rate of Valsalva manoeuvre with device to supraventricular tachycardia was 50%. We powered our study to be able to detect at least a 20% absolute improvement with the modified Valsalva manoeuvre, using the available evidence and the minimum improvement we thought would effect a change in practice. We estimated that this difference would require 106 patients per group (assuming a two-tailed test of statistical significance with an α of 0·05 and power of 0·9), and a 12 months recruitment period in our center.

- Statistical Analysis: Participants were analysed according to intention to treat, and endpoints will be attributed to the treatment arm to which the patients were randomized, regardless of treatment crossover or post-randomization medical care. The statistical analysis will be carried out in accordance with the pre-designed. We compared binary outcomes (including the primary outcome and the secondary outcome) using mixed effects logistic regression with allocation group as a fixed effect and clinicians as a random effect.

ELIGIBILITY:
Inclusion Criteria:

* Patient having supraventricular tachycardia (SVT) with regular, narrow complex tachy-arrythmia with a QRS duration < 0.12 ms on ECG and eligible for treatment with the Valsalva manoeuvre.
* AVNRT (atrioventricular nodal re-entry tachycardia) or AVRT (atrioventricular re-entry tachycardia) conformed by electrophysiologic test.

Exclusion Criteria:

* Unable or unwilling to give informed verbal consent.
* SVT episode with hemodynamic instability (systolic blood pressure (BP) < 90 mmHg).
* With atrial fibrillation or atrial flutter.
* Severe hypertension (systolic BP > 220 mmHg or diastolic BP > 120 mmHg).
* Contraindication or inability to perform a VM (aortic stenosis, recent myocardial infarction, glaucoma, retinopathy, recent eye surgery, paralysis).
* Third trimester pregnancy.
* Previous catheter ablation of SVT.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
The presence of sinus rhythm | From enrollment to the end of treatment at 1 day.
  The primary outcome is the presence of sinus rhythm as recorded by the treating clinician 1 min after twice VM and confirmed by ECG in the intention-to-treat population.

SECONDARY OUTCOMES:
The presence of sinus rhythm | From enrollment to the end of treatment at 1day
  Secondary outcomes are the presence of sinus rhythm as recorded by the treating clinician 1 min after once VM, and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Songnan Li, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Capital Medical University affiliated Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 6 months after the publication of results.
Access Criteria: A proposal that describes planned analyses must be submitted and a data sharing agreement must be signed. And the plan must be approved by Dr. Songnan Li.

REFERENCES:
- [Derived] Huang L, Sang C, Gao M, Lai Y, Zhang J, Wang Y, Guo L, Liu N, Liu X, Guo X, Guo Q, Zuo S, Li C, Jiang C, Zhao Z, Tang R, Li S, Long D, Du X, Dong J, Ma C, Macle L. Device-Assisted vs Standard Valsalva Maneuver for Terminating Supraventricular Tachycardia: A Randomized Clinical Trial. JAMA Cardiol. 2026 Feb 11. doi: 10.1001/jamacardio.2025.5489. Online ahead of print. PMID 41670992